CLINICAL TRIAL: NCT03052673
Title: Per-operative Low-Dose Ketamine For Postoperative Pain Relief In Patients Undergoing Bariatric Surgery: A Randomised Study
Brief Title: Ketamine for Pain Relief in Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Dr Nitin Sethi, Doctor & Associate Professor, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC/01/17/1120
Record Dates: First submitted 2017-02-06; First posted 2017-02-14 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Pain
Keywords: ketamine; fentanyl; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Ketamine

STUDY DESIGN:
Intervention Model Description: 76 patients belonging to ASA physical patients status II and III of either sex, scheduled to undergo laparoscopic bariatric surgery (sleeve gastrectomy, Roux-en-Y gastric bypass) under general anaesthesia. The patients will be randomly allocated by computer generated numbers to one of the following two groups of 38 patients each.
  Group 1[Ketamine + Fentanyl Group, n=38]: Pre-induction fentanyl 1-mcg/kg, ketamine 0.5-mg/kg after induction, followed by intraoperative fentanyl infusion of 0.5-mcg/kg/hr + ketamine infusion of 0.2-mg/kg/hr.
  Group 2[Fentanyl Group, n=38]:Pre-induction fentanyl 1-mcg/kg, saline after induction followed by intraoperative fentanyl infusion of 0.5-mcg/kg/hr + saline infusion.
  Both the groups will receive intravenous PCA of fentanyl post-operatively
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient and the attending anaesthesiologist will be blinded to the intraoperative infusions used. Postoperative patient recovery profile will also be evaluated by an independent assess or blinded to the intraoperative anaesthesia technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine + Fentanyl Group (Active Comparator): Patients will receive pre-induction fentanyl 1-mcg/kg, ketamine 0.5-mg/kg after induction, followed by intraoperative fentanyl infusion of 0.5-mcg/kg/hr + ketamine infusion of 0.2-mg/kg/hr.
  Postoperative analgesia will be provided with Intravenous Patient Controlled Analgesia (IV-PCA) pump containing fentanyl citrate-2.5 mcg/ml, which will be attached to all the patients upon shifting to the recovery room. The IV-PCA pump settings will be as follows: 0-ml basal dose; 4-ml PCA dose; 15-minutes lock out interval.
  Interventions: Drug: Fentanyl; Drug: ketamine
- Fentanyl Group (Active Comparator): Patients will receive pre-induction fentanyl 1-mcg/kg,followed by intraoperative fentanyl infusion of 0.5-mcg/kg/hr.
  Postoperative analgesia will be provided with Intravenous Patient Controlled Analgesia (IV-PCA) pump containing fentanyl citrate-2.5 mcg/ml, which will be attached to all the patients upon shifting to the recovery room. The IV-PCA pump settings will be as follows: 0-ml basal dose; 4-ml PCA dose; 15-minutes lock out interval.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl 1mcg/kg will be given at induction of anaesthesia followed by intraoperative infusion of 0.5 mcg/kg/hr in both the arms . Postoperatively IV-PCA pump containing fentanyl will be attached to patients in both the arms
Drug: ketamine — Ketamine 0.5 mg/kg will be given post-induction of anaesthesia followed by infusion of 0.5 mcg/kg /hr in the Ketamine + Fentanyl group arm
  Arms: Ketamine + Fentanyl Group

SUMMARY:
The surgical interventions for treating morbid obesity, i.e. bypass procedure and sleeve gastrectomy are collectively covered under the term 'bariatric surgery'. The growth of bariatric surgery has seen consonant development of anaesthesia techniques so as to ensure patient safety and facilitate post-surgery outcome. Conventionally, balanced general anaesthesia techniques routinely use opioids peri-operatively for intra-operative haemodynamic homeostasis and postoperative pain relief. However, since the morbidly obese patients have high prevalence of obstructive sleep apnea(OSA) and other co-morbidities the same technique when employed in the morbidly obese patients hampers early and intermediate postoperative recovery due to the occurrence of side effects, such as, sedation, PONV, respiratory depression, depressed GI-mobility. The above stated side effects, have lead to increased propensity for postoperative cardiac and pulmonary complications. Obese patients are more vulnerable and sensitive to the narcotics and sedatives, these drugs need to be employed judiciously in these patients. On the other hand, the reduction in opioid use may result in acute post-operative pain that may limit post-surgery rehabilitation. Therefore, we need to minimise opioid use and employ some other drugs which besides having analgesia, has a opioid-sparing effect also.

Ketamine, an N-methyl-D-aspartate (NMDA) receptor antagonist, has analgesic properties in sub-anaesthetic doses. When used in low dose (0.2mg/kg), it is an analgesic, anti-hyperalgesic, and prevents development of opioid tolerance. On a conceptual basis, a key advantage of ketamine is that it can reduces post-operative pain and use of opioid when used per-operatively. Therefore, a regimen which avoid or minimise use of opioid is likely to decrease opioid-related postoperative morbidity in these patients undergoing bariatric surgery.In view of the above, a clinical research is highly desirable to study techniques to decrease the use of opioids in obese surgical patients.This prospective randomised two-arm study aims to assess the effect of low-dose ketamine on postoperative pain relief and opioid-sparing ability in obese patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
After obtaining approval from the hospital ethics committee and written informed consent from the patients, this prospective randomised study will be conducted on 76 patients belonging to ASA physical patients status II and III of either sex, scheduled to undergo laparoscopic bariatric surgery (sleeve gastrectomy, Roux-en-Y gastric bypass) under general anaesthesia. The patients will be randomly allocated by computer generated numbers to one of the following two groups of 38 patients each.

Group 1[Ketamine + Fentanyl Group, n=38]: Pre-induction fentanyl 1-mcg/kg, ketamine 0.5-mg/kg after induction, followed by intra-operative fentanyl infusion of 0.5-mcg/kg/hr + ketamine infusion of 0.2-mg/kg/hr

Group 2[Fentanyl Group, n=38]: Pre-induction fentanyl 1-mcg/kg, saline after induction followed by intra-operative fentanyl infusion of 0.5-mcg/kg/hr + saline infusion.

Both the groups will receive intravenous PCA of fentanyl post-operatively.

Randomisation, Allocation Concealment:

The patients will be randomly allocated to one of the two groups based on a computer-generated random number table (url:stattrek.com/statistics/random-number-generator.aspx). Randomisation sequence concealment will include opaque-sealed envelopes with alphabetic codes whose distribution will be in control of an independent analyst. The envelopes will be opened; patient's data-slip will be pasted on them, and will be sent back to the control analyst.

Blinding Strategy:

The attending anaesthesiologist will be blinded to the intra-operative infusions used. Postoperative patient recovery profile will also be evaluated by an independent assess or blinded to the intra-operative anaesthesia technique.

Management of Anaesthesia:

Premedication

All patients will be receive tablet ranitidine-150 mg night before and on morning of surgery.They will be instructed to fast for at least 8- hours before surgery. Clear fluids will be allowed till 2 hours before surgery.

Intra-operative Monitoring

Two peripheral venous lines (18G/20G catheter) will be secured. Standard monitoring including 5-lead ECG, non-invasive blood pressure (NIBP), pulse oximeter, end-tidal carbon dioxide (EtCO2) and end-tidal gas monitoring will be applied. Additional monitoring will include depth of anaesthesia monitoring using Bi-spectral index (BIS) and neuromuscular monitoring using train-of-four response.

Anaesthesia Technique

All patients will be pre-oxygenated with 100% oxygen for at least 3-minutes prior to induction of anaesthesia. All the drugs (study + control) will be administered based on lean body weight (LBW). Patients in the KF group will receive pre-induction fentanyl-citrate l-µg/kg IV and ketamine 0.5-mg/kg after induction whereas patients in the Fentanyl group will receive pre-induction fentanyl-citrate l-µg/kg IV and saline as in above group. Anaesthesia will be induced with propofol 2-2.5mg/kg titrated to a BIS-value of 50.. After induction of anaesthesia, atracurium besylate 0.5-mg/kg will be administered for skeletal muscle relaxation to facilitate tracheal intubation. Ventilator settings for CMV, tracheal tube size [7.5-mm I.D (male), 6.5-mm I.D (female)], and breathing circuit (circle-CO2 absorber system) will be the standardised in all the patients. The patients in the Ketamine + Fentanyl group will receive fentanyl infusion at 0.5-mcg/kg/hr and ketamine infusion of 0.2-mg/kg/hr. The patients in the Fentanyl group will receive fentanyl infusion at 0.5-mcg/kg/hr and saline infusion. The LBW in obesity patients scheduled to undergo bariatric surgery will be calculated based on the following formulae:

9270 x TBW (kg)/6680 + (216 x BMI) [men]

9270 x TBW (kg)/8780 + (244 x BMI) [women]

Desflurane in oxygen-nitruos oxide mixture (FiO2 0.50) will be used for maintenance in both the groups to maintain a BIS of 40-60. Intra-operative muscle relaxation will be maintained using atracurium boluses controlled by train-of-four response on peripheral neuromuscular monitor. Thirty minutes before the end of surgery, non-opioid analgesics, such as paracetamol 1-gm will be administered to the patient. Desflurane delivery will be stopped at the point of completion of skin closure. Residual neuromuscular blockade (assessed with train-of-four response) will be reversed with neostigmine (50-µg/kg) and glycopyrrolate (20-µg/kg).

After discontinuation of anaesthesia delivery (0-time point) the time to eye opening and time to extubation will be determined. After tracheal extubation the patients will be shifted to postoperative recovery room adjoining OT suites and will be closely observed for oxygenation and ventilation status, pain (visual analogue score [VAS]), sedation (Modified OASS), and PONV.

Intravenous Patient Controlled Analgesia (IV-PCA) pump containing fentanyl citrate-2.5 mcg/ml will be attached to all the patients upon shifting to the recovery room. The IV-PCA pump settings will be as follows: 0-ml basal dose; 4-ml PCA dose; 15-minutes lock out interval. A baseline visual analogue scoring will be done after shifting the patient to the recovery room (0-time point) followed by 2-hours, 4-hours, 8-hours, 12-hours, and 24-hours time points from the baseline. Any adverse effects such as hypotension/ hypertension, bradycardia/tachycardia, hypoxemia, giddiness will be recorded and treated. Post-surgery, time to alimentation post surgery will be noted.

'Rescue' pain relief drug will include: diclofenac sodium 75 mg slow IV bolus for NRS>3 and 'rescue' antiemesis agent would be ondansetron 4-mg for a PONV score > 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 18-60 years
* BMI > 35 kg/m2
* Either sex
* ASA physical status II & III
* undergoing laparoscopic bariatric surgery

Exclusion Criteria:

* Patients refusal
* ASA physical status: IV
* History of hypersensitivity to fentanyl and/or ketamine
* Chronic opioid use
* History of substance abuse
* Metabolic disorders
* Seizure disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of Postoperative Analgesia | From end of anaesthesia till 24-hours postoperatively
  will be assessed using visual analogue scale (VAS) score
Postoperative Fentanyl Consumption in micrograms | From end of anaesthesia till 24-hours postoperatively
  Amount of fentanyl consumed using the IV-PCA pump will be calculated

SECONDARY OUTCOMES:
Time to eye opening in minutes | From end of anaesthesia till 20-minutes postoperatively
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Time to extubation in minutes | From end of anaesthesia till 30-minutes postoperatively
  Time taken for tracheal extubation after discontinuation of anaesthesia will be noted
Changes in intraoperative heart rate (beats per minute) | From beginning of anesthesia (0-hours, baseline) till 6 hours intraoperatively
  Comparison of intraoperative heart rate between both the arms will be done
Changes in intraoperative blood pressure- systolic, diastolic, and mean (mmHg) | From beginning of anesthesia (0-hours, baseline) till 6 hours intraoperatively
  Comparison of intraoperative blood pressure- systolic, diastolic, and mean between both the arms will be done
Postoperative Sedation | From end of anaesthesia till 24-hours postoperatively
  will be assessed using Modified Observer's assessment of alertness/sedation scale (OASS)
Postoperative Nausea and Vomiting | From end of anaesthesia till 24-hours postoperatively
  will be assessed using PONV Scale

CONTACTS AND LOCATIONS:
Overall Officials: Haider Hussain, MBBS, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA; Anil K Jain, MD, Study Chair — Sir Ganga Ram Hospital, New Delhi, INDIA; Amitabh Dutta, MD, Study Director — Sir Ganga Ram Hospital, New Delhi, INDIA; Nitin Sethi, DNB, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA; Praveen Bhatia, MS, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, India

IPD SHARING:
Plan to Share IPD: No